CLINICAL TRIAL: NCT04003987
Title: Erector Spinae Plane Block Versus Transverse Abdominis Plane Block in Laparoscopic Hysterectomy
Brief Title: ESP Block VS TAP in Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Yar Yeap, Director, Acute Pain Service Assistant Professor of Clinical Anesthesiololgy Department of Anesthesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1903977303
Record Dates: First submitted 2019-05-23; First posted 2019-07-01 (Actual); Results first posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Hysterectomy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: 1. ESP Block Group
  2. TAP Block Group
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the patients and the research staff doing assessments will be blinded to the randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ESP Block (Active Comparator): For the ESP block the ultrasound is positioned in a parasagittal fashion, 2-3 inches lateral to the spinous process. This approach visualizes the transverse process. The needle is inserted cranial-to-caudal to make contact with the shadow of the transverse process, with the needle tip deep to the fascial plane of the erector spinae muscle. Injection of saline confirms the location of the needle, and the anesthetic is injected (40 ml into each side; 20 ml injected at T8 and 20 ml injected at T12)
  Interventions: Drug: Liposomal bupivacaine; Drug: bupivacaine, 0.125%
- TAP Block (Active Comparator): For the TAP block, the ultrasound probe is placed transverse to the abdominal wall, between the iliac crest and the costal margin. The needle is placed in the plane of the probe and advanced until it is between the internal oblique and the transversus abdominis muscles. Once in the plane, 2 mL of saline is injected to confirm needle position, then the local anesthetic solution is injected (40 ml into each side; 20 ml injected for subcostal TAP and 20 ml injected for posterior TAP).
  Interventions: Drug: Liposomal bupivacaine; Drug: bupivacaine, 0.125%

INTERVENTIONS:
Drug: Liposomal bupivacaine — 20ml
  Other Names: Exparel
Drug: bupivacaine, 0.125% — 60ml
  Other Names: bupivacaine

SUMMARY:
The purpose of this study is to compare the difference between two different pain control methods in patients who will be having a hysterectomy surgery. By collecting this data, we aim to show improved postoperative pain scores, decreased opioid needs, and decreased opioid side effects (nausea, sedation, ileus, urinary retention, respiratory depression).

DETAILED DESCRIPTION:
For the TAP block, the ultrasound probe is placed transverse to the abdominal wall, between the iliac crest and the costal margin. The needle is placed in the plane of the probe and advanced until it is between the internal oblique and the transversus abdominis muscles. Once in the plane, 2 mL of saline is injected to confirm needle position, then the local anesthetic solution is injected. [10]

For the ESP block, as mentioned previously, the ultrasound is positioned in a parasagittal fashion, 2-3 inches lateral to the spinous process. This approach visualizes the transverse process. The needle is inserted cranial-to-caudal to make contact with the shadow of the transverse process, with the needle tip deep to the fascial plane of the erector spinae muscle. Injection of saline confirms the location of the needle, and the anesthetic is injected.

All patients will receive PO acetaminophen and PO gabapentin the morning of surgery. Pt. will be placed on PRN oxycodone/acetaminophen (Percocet) postoperatively. PRN IV dilaudid may be given for severe breakthrough pain.

Opioid usage at 1, 24 and 48 hours after the block will be recorded by a member of the research team. Pain scores at rest and on movement will be measured by the investigator using Visual Analog Scale (VAS). Nausea will be measured using a categorical scoring system (none=0; mild=1; moderate=2; severe=3). Sedation scores will also be assessed by a member of the study team using a sedation scale (awake and alert=0; quietly awake=1; asleep but easily roused=2; deep sleep=3). All these parameters will be measured at 1, 24 and 48 hours after the blocks and patients will be encouraged to ambulate on postoperative day 1 under supervision. Their ambulation activity will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic hysterectomy surgery at Indiana University Hospital
* ASA class 1, 2, 3 or 4
* Age 18 or older, female
* Desires Regional anesthesia for postoperative pain control

Exclusion Criteria:

* History of substance abuse in the past 6 months.
* Patients on more than 30 mg morphine equivalents of opioids.
* Any physical, mental or medical conditions which in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery.
* Known allergy or other contraindications to the study medications (Acetaminophen, Gabapentin, Bupivacaine).
* Postoperative intubation.
* Any BMI greater than 40.0.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yar Yeap, MD, Principal Investigator — Indiana University Hospital; Matthew Warner, MD, Principal Investigator — Indiana University Hospital
Locations (2):
- United States (2):
  - Indiana Univeristy, Indianapolis, Indiana
  - Indiana University Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shaffer EE, Pham A, Woldman RL, Spiegelman A, Strassels SA, Wan GJ, Zimmerman T. Estimating the Effect of Intravenous Acetaminophen for Postoperative Pain Management on Length of Stay and Inpatient Hospital Costs. Adv Ther. 2017 Jan;33(12):2211-2228. doi: 10.1007/s12325-016-0438-y. Epub 2016 Nov 9. PMID 27830448
- [Result] Routman HD, Israel LR, Moor MA, Boltuch AD. Local injection of liposomal bupivacaine combined with intravenous dexamethasone reduces postoperative pain and hospital stay after shoulder arthroplasty. J Shoulder Elbow Surg. 2017 Apr;26(4):641-647. doi: 10.1016/j.jse.2016.09.033. Epub 2016 Nov 15. PMID 27856266
- [Result] Bacal V, Rana U, McIsaac DI, Chen I. Transversus Abdominis Plane Block for Post Hysterectomy Pain: A Systematic Review and Meta-Analysis. J Minim Invasive Gynecol. 2019 Jan;26(1):40-52. doi: 10.1016/j.jmig.2018.04.020. Epub 2018 Apr 30. PMID 29723644
- [Result] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Result] Petsas D, Pogiatzi V, Galatidis T, Drogouti M, Sofianou I, Michail A, Chatzis I, Donas G. Erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: a case report. J Pain Res. 2018 Sep 24;11:1983-1990. doi: 10.2147/JPR.S164489. eCollection 2018. PMID 30288093
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Vyas KS, Rajendran S, Morrison SD, Shakir A, Mardini S, Lemaine V, Nahabedian MY, Baker SB, Rinker BD, Vasconez HC. Systematic Review of Liposomal Bupivacaine (Exparel) for Postoperative Analgesia. Plast Reconstr Surg. 2016 Oct;138(4):748e-756e. doi: 10.1097/PRS.0000000000002547. PMID 27673545
- [Result] Hadzic A, Minkowitz HS, Melson TI, Berkowitz R, Uskova A, Ringold F, Lookabaugh J, Ilfeld BM. Liposome Bupivacaine Femoral Nerve Block for Postsurgical Analgesia after Total Knee Arthroplasty. Anesthesiology. 2016 Jun;124(6):1372-83. doi: 10.1097/ALN.0000000000001117. PMID 27035853
- [Result] Wu ZQ, Min JK, Wang D, Yuan YJ, Li H. Liposome bupivacaine for pain control after total knee arthroplasty: a meta-analysis. J Orthop Surg Res. 2016 Jul 22;11(1):84. doi: 10.1186/s13018-016-0420-z. PMID 27443874
- [Derived] Warner M, Yeap YL, Rigueiro G, Zhang P, Kasper K. Erector spinae plane block versus transversus abdominis plane block in laparoscopic hysterectomy. Pain Manag. 2022 Nov;12(8):907-916. doi: 10.2217/pmt-2022-0037. Epub 2022 Oct 10. PMID 36214314

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ESP Block | TAP Block
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESP Block | TAP Block | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 39 | 78
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (1.9) | 42.7 (1.8) | 44.9 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) Pain Scores at Rest at 1 Hour.
Description: Visual Analogue Scale (VAS) score taken at rest is measured as minimal to maximal; higher values mean worse pain (scale 0-10)
Time Frame: 1 hour after surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 39 | 39
score on a scale | 2.8 (0.5) | 3 (0.4)

2. Primary Outcome: Visual Analogue Scale (VAS) Pain Scores at Rest at 24 Hours.
Description: Visual Analogue Scale (VAS) score taken at rest measured as minimal to maximal; higher values mean worse pain (scale 0-10)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 39 | 39
score on a scale | 3 (0.4) | 2.8 (0.4)

3. Primary Outcome: Visual Analogue Scale (VAS) Pain Scores at Rest at 48 Hours.
Description: Visual Analogue Scale (VAS) score taken at rest measured as minimal to maximal; higher values mean worse pain(scale 0-10)
Time Frame: 48 hours after surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 39 | 39
score on a scale | 2.1 (0.4) | 2 (0.3)

4. Primary Outcome: Visual Analogue Scale (VAS) Pain Scores With Movement at 1 Hour.
Description: Visual Analogue Scale (VAS) score taken with movement is measured as minimal to maximal; higher values mean worse pain (scale 0-10)
Time Frame: 1 hour after surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 39 | 39
score on a scale | 3 (0.5) | 3.5 (0.4)

5. Primary Outcome: Visual Analogue Scale (VAS) Pain Scores With Movement at 24 Hours.
Description: Visual Analogue Scale (VAS) score taken with movement measured as minimal to maximal; higher values mean worse pain (scale 0-10)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 39 | 39
score on a scale | 4.3 (0.4) | 4.1 (0.4)

6. Primary Outcome: Visual Analogue Scale (VAS) Pain Scores With Movement at 48 Hours.
Description: Visual Analogue Scale (VAS) score taken with movement measured as minimal to maximal; higher values mean worse pain(scale 0-10)
Time Frame: 48 hours after surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 39 | 39
score on a scale | 3.4 (0.4) | 3.2 (0.3)

7. Secondary Outcome: Patient Sedation Score at 1 Hour
Description: Sedation is measured as minimum to maximum awareness/level of consciousness; higher values means worse or less awareness (awake, asleep but arousable, deep sleep)
Time Frame: 1 hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 38 | 39
Participants
  Sleep | 15 | 15
  Awake | 23 | 24

8. Secondary Outcome: Patient Sedation Score at 24 Hours
Description: Sedation is measured as minimum to maximum aware ness/level of consciousness: higher values means worse or less awareness (awake, asleep but arousable, deep sleep)
Time Frame: 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 36 | 39
Participants
  Sleep | 2 | 1
  Awake | 34 | 38

9. Secondary Outcome: Patient Sedation Score at 48 Hours
Description: as for outcome 7
Time Frame: 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 35 | 39
Participants
  Sleep | 0 | 1
  Awake | 35 | 38

10. Secondary Outcome: Patient Nausea Score at 1 Hour
Description: Nausea is measured as minimum to maximum: higher values is worse (none, mild, moderate, severe)
Time Frame: 1 hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 38 | 39
Participants
  Yes | 5 | 6
  No | 33 | 33

11. Secondary Outcome: Patient Nausea Score at 24 Hour
Description: Nausea is measured as minimum to maximum: higher values is worse (none, mild, moderate, severe)
Time Frame: 24 hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 36 | 39
Participants
  Yes | 11 | 7
  No | 25 | 32

12. Secondary Outcome: Patient Nausea Score at 48 Hour
Description: Nausea is measured as minimum to maximum: higher values is worse (none, mild, moderate, severe)
Time Frame: 48 hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 35 | 39
Participants
  Yes | 2 | 7
  No | 33 | 32

13. Secondary Outcome: Patient Satisfaction Score at 24 Hours
Description: patient satisfaction is measured as minimum to maximum 1-5; the higher the score the better satisfied (very unsatisfied, unsatisfied, neutral, satisfied, very satisfied)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 36 | 39
score on a scale | 3.7 (0.1) | 3.6 (0.1)

14. Secondary Outcome: Patient Satisfaction Score at 48 Hours
Description: as for outcome 13
Time Frame: 48 hours after surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ESP Block | TAP Block
Number analyzed (Participants) | 36 | 39
score on a scale | 3.7 (0.1) | 3.7 (0.1)

ADVERSE EVENTS:
Time Frame: From the time of consent up to 6 months after surgery.
Arm/Group | ESP Block | TAP Block
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04003987/Prot_SAP_000.pdf